CLINICAL TRIAL: NCT04401969
Title: Studying the Tissue Microenvironment Signatures of the Mycetoma Granuloma
Brief Title: Tissue Microenvironment Signatures of the Mycetoma Granuloma
Status: Completed | Type: Observational
Sponsor: University of Khartoum (Other)
Collaborators: University of York (Other)
Responsible Party: Principal Investigator, Dr Mohamed Osman, Principal Investigator, University of Khartoum
Other Study IDs: Mycetoma Study
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Mycetoma
MeSH Terms: conditions — Mycetoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Needle biopsy samples from mycetoma lesions
  Fine needle aspirates from the matching mycetoma lesion
  Whole blood for RNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with eumycetoma lesions: Patients with eumycetoma lesions
- Patients with actinomycetoma lesions: Patients with actinomycetoma lesions
- Patients with lesions of unknown causality: Patients with lesions of unknown causality

SUMMARY:
Mycetoma is the most neglected of the neglected tropical diseases. It is caused by certain fungi or bacteria. It is endemic in many tropical and subtropical regions and Sudan seems to be the mycetoma homeland. This chronic subcutaneous destructive and disabling inflammatory disease has many serious medical and socio-economic impacts on patients, community and health authorities. This work may suggest new therapeutic options for mycetoma that target the inflammatory pathogenic pathway and hence help in designing universal treatment options for mycetoma patients.

Two overlapping aims were investigated in this project to advance our overall goals:

1. Profiling the immune/inflammatory signatures in the tissue microenvironment of fungus-induced mycetoma lesions
2. Profiling the immune/inflammatory signatures in the tissue microenvironment of bacteria-induced mycetoma lesions.

DETAILED DESCRIPTION:
Mycetoma is a chronic, specific, subcutaneous granulomatous, progressive and disfiguring inflammatory disease. It is caused by true fungi or by certain bacteria and hence it is usually classified into eumycetoma and actinomycetoma respectively. Madurella mycetomatis is the commonest eumycetoma causative agent, while Streptomyces somaliensis and Nocardia brasiliensis are the common causative organisms for actinomycetoma. The triad of a painless subcutaneous mass, sinuses formation and purulent or sero-purulent discharge that contains grains is pathognomonic of mycetoma. The inflammatory subcutaneous granuloma usually spreads to involve the skin and the deep structures, resulting in destruction, deformity and loss of function, occasionally it can be fatal. The foot and hand are the most frequently affected sites seen in 82% of cases. In endemic areas, other parts of the body may be involved such as the knee, arm, leg, head and neck, thigh and perineum. No age is exempted in mycetoma; however, it occurs more frequently in young adult men in the age range 20-40 years and almost 30% of reported patients were young students.

The true incidence and prevalence of mycetoma world-wide is not precisely known. It is interesting to note that most of the reported mycetoma data are related to hospital patients with advanced disease. This is attributed to the nature of mycetoma which is usually painless, slowly progressive and the late presentation of the majority of patients due to the poor health education, lack of health facilities and financial constraints.

The worldwide distribution of mycetoma varies widely. It is endemic in many tropical and subtropical regions and prevails in the mycetoma belt, which includes the countries of Sudan, Somalia, Senegal, India, Yemen, Mexico, Venezuela, Columbia, Argentina, and a few others. The African continent seems to have the highest burden and prevalence of the disease. It has also been extensively reported from India. However, mycetoma has been reported in many temperate regions as well. There are a few reports on mycetoma from the USA, Sri Lanka, Germany, Egypt, Turkey, Philippines, Japan, Lebanon, Thailand, Saudi Arabia, Tunisia and Iran.

The proper treatment of mycetoma depends mainly on accurate diagnosis. It is essential to identify the causative organism to the species level and the current tests for that are the classical grains culture, surgical biopsy histopathological examination and various molecular techniques such as PCR. Various imaging techniques such as conventional radiology, ultrasonography, CT scan and MRI are in use to determine the disease extend. Most of these tests and techniques are invasive, expensive and of low sensitivity and specificity. Furthermore, they are not available in the mycetoma endemic regions and hence there is a desperate need forth easy to use, field-friendly test to identify the causative agent.

The management of this distressing and devastating disease is disappointing. The treatment depends mainly on the aetiological agent, the site and extend of the disease. Until recently, the only available treatment for mycetoma was amputation or multiple mutilating disfiguring surgical excisions. Combined medical treatment in the form of antifungals for the eumycetoma and antibiotics and antimicrobial agents for actinomycetoma and various surgical excisions is the gold standard in mycetoma.

Reports on medical treatment in eumycetoma are scarce and inadequate. Over the years and till now, the treatment of eumycetoma was based on personal clinical experience and on the results of sporadic case reports, rather than controlled clinical trials. In general, massive surgical excisions or amputation of affected part is the treatment of choice for eumycetoma. Various antifungal agents have been tried with little success. This is perhaps surprising, as the eumycetoma causative agents are low-grade infective organisms and their eradication should be readily achieved by the administration of antifungal drugs. Generally, actinomycetoma is amenable to medical treatment with antibiotics and other chemotherapeutic agents. Combined drug therapy is always preferred to a single drug to avoid drug resistance and for disease eradication.

Medical treatment for both types of mycetoma must continue until the patient is clinically, radiologically, ultrasonically and cytologically cured. Recurrence is more common after an incomplete or irregular course of medical treatment. With patient non-compliance, there is a good chance for the organism to develop drug resistance.

The study was conducted at the Mycetoma clinic at the Mycetoma Research Centre (MRC), Khartoum Sudan. Patients were enrolled into the study after written informed consent was obtained in line with the Declaration of Helsinki.

Patients were categorized into three groups;

* Patients with eumycetoma lesions (n=10)
* Patients with actinomycetoma lesions (n=12)
* Patients with lesions of unknown causality (n=6)

Formalin fixation and paraffin embedding was performed at the MRC according to standard procedures.

Fine needle aspirates (FNA) was collected for flow cytometry at the same time and at the same location of the lesion in the body.

Aspirates were frozen at -80C for future analysis. Concurrently, 15 ml of blood was taken from each patient for immunological function assays.

Peripheral blood mononuclear cells were prepared using standard protocols and stored in liquid nitrogen till required.

5 ml of blood was collected in Paxgene tubes for transcriptomics analysis.

Immunohistochemistry Immunohistochemistry was performed at University of York, UK. Formalin fixed paraffin embedded (FFPE) sections were analysed using the 700 gene Nanostring PanCancer Immune Cell profiling panel to obtain a high level view of the immune/inflammatory signature.

Serial sections were subjected to highly multiplexed antibody staining using the Nanostring Digital Spatial Profiling system to obtain a comprehensive and spatially resolved insights into lesion microenvironment.

Candidate pan-mycetoma targets identified by these approaches were confirmed using immunofluorescent antibodies and RNA-fluorescent in situ hybridisation.

All data was recorded as digitised whole slide images for publication and archiving.

Antigen specific T cell responses T cells responses analysis were performed at Institute for Endemic Diseases, University of Khartoum.

Peripheral blood mononuclear cells (PBMCs) from patients and age and sex matched healthy control from endemic area were stimulated for 7 days with fungus and bacterial lysates. IFN, IL-17, IL-4 and IL-10 responses were determined by ELISPOT assay.

Flow cytometry on FNBs were performed with panels of antibodies to evaluate T cell and myeloid cell phenotype.

Whole blood transcriptomics Blood were collected into Paxgene and stored at - 80c. RNA were extracted from stored samples Full whole blood transcriptomic data was obtained by RNA-Seq.

Cytokine measurements in mycetoma aspirates were undertaken using commercially available ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

Patients aged over 18 years with either small or advanced eumycetoma lesions with either small or advanced actinmycetoma lesions with lesions of unknown causality

Exclusion Criteria:

<18 years of age Inability to provide informed consent Any other reason that in the opinion of the Investigator indicates the subject cannot comply with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from Soba University Hospital Mycetoma clinic
  10 patients with eumycetoma lesions 12 patients with actinomycetoma lesions 6 patients with lesions of unknown causality
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
immune cell phenotypes | 24 months
  detection of immune cell phenotypes in mycetoma lesions
antigen-specific t-cell responses | 24 months
  detection of t cell and myeloid cell phenotype in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Osman, PhD, Principal Investigator — University of Khartoum
Locations (1):
- University Hospital Soba, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: No